CLINICAL TRIAL: NCT00176215
Title: Clinical Comparison of RPDs Retained by Conical and Galvanoformed Double Crowns.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG-FL-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Denture, Partial, Removable; Dental Prosthesis Retention; Oral Health; Tooth Abrasion
MeSH Terms: conditions — Tooth Abrasion

INTERVENTIONS:
Procedure: survival failure of more than 20 %

SUMMARY:
The aim of this prospective clinical trial was to investigate the clinical performance and complication rate of RPDs (Removable partial dentures) retained on conventional conical double crowns in comparison to galvanoformed telscopic double crowns. Additionally the OHIP (Oral Health related Qualitiy of Life)and the abrasion of the teeth were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Indication for RPDs retained by double crowns; 2 to 6 Abutment teeth;

Exclusion Criteria:

* limited contractual capability and absence of consent of the patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Grossmann, DDS, Study Chair — Heidelberg University; Franziska Lehmann, DDS, Principal Investigator — Heidelberg University
Locations (2):
- Germany (2):
  - University of Heidelberg, Heidelberg, Baden-Wurttemberg
  - University of Heidelberg, Heidelberg, Baden_Württemberg